CLINICAL TRIAL: NCT07274410
Title: Clinical Profile And Outcome Of Neonatal Convulsions Among Newborns Admitted To The Neonatal Intensive Care Unit At Assiut University Children's Hospital: A Prospective Cohort Study
Brief Title: Clinical Profile And Outcomes Of Neonatal Convulsions In The Neonatal Intensive Care Unit At Assiut University Children's Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, zeinab ahmed abdel sabour, Resident, Pediatrics, Assiut University
Other Study IDs: NC-ASSIUT-2024
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Neonatal Convulsions; Newborn Seizure Disorders; Seizures
Keywords: Neonatal convulsions; Neonatal ICU; outcomes
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonatal Convulsions: This cohort includes neonates aged 0-30 days who are admitted to the Neonatal Intensive Care Unit at Assiut University Children's Hospital and diagnosed with neonatal convulsions. Participants will undergo clinical evaluation, laboratory investigations, neuroimaging, and follow-up to assess seizure characteristics, underlying etiologies, management, and outcomes. No interventions will be assigned; only observational data will be collected.
  Interventions: Other: Management of Neonatal Convulsions

INTERVENTIONS:
Other: Management of Neonatal Convulsions — This intervention involves the clinical management of neonatal convulsions in newborns aged 0-30 days admitted to the NICU. Management includes prompt identification of seizure activity through clinical evaluation and EEG confirmation, followed by appropriate treatment using anticonvulsant medications such as phenobarbital. Supportive care includes monitoring of vital signs, glucose, and electrolytes, and performing necessary investigations like abdominal ultrasound, echocardiography, and brain imaging (MRI/CT) to identify underlying causes. The intervention aims to control seizures, minimize neurological complications, and improve short-term and long-term outcomes in affected neonates.

SUMMARY:
Neonatal convulsions are seizures that occur during the first 28 days of a newborn's life. They are considered a medical emergency and often indicate an underlying problem in the brain, such as lack of oxygen at birth, infections, metabolic disturbances, or structural abnormalities. Many seizures in newborns are subtle and difficult to detect without careful clinical assessment.

This study aims to determine how often neonatal convulsions occur among newborns admitted to the Neonatal Intensive Care Unit (NICU) at Assiut University Children Hospital. It will describe how affected newborns present clinically, identify the main causes, and evaluate the early outcomes during hospitalization.

The study is designed as a prospective cohort study. Newborns aged 0-30 days who are diagnosed with neonatal convulsions will be enrolled and followed throughout their stay in the NICU. Each patient will undergo full clinical evaluation and standard laboratory and imaging investigations, including blood tests, neuroimaging, and other tests as clinically indicated.

The findings of this study will provide updated local data on the incidence, causes, and outcomes of neonatal convulsions in our region. This information may help improve early diagnosis, guide appropriate treatment, and enhance the quality of neonatal care.

DETAILED DESCRIPTION:
Neonatal convulsions represent one of the most important neurological emergencies in early life and are strongly associated with underlying brain dysfunction. In many cases, the clinical manifestations are subtle, making diagnosis challenging without careful observation and appropriate diagnostic tools. Early recognition of neonatal seizures and identification of their etiologies play essential roles in preventing long-term neurological complications.

This prospective cohort study is designed to investigate the clinical profile and outcomes of neonatal convulsions among newborns admitted to the Neonatal Intensive Care Unit at Assiut University Children Hospital. The study will include newborns aged 0 to 30 days, of both sexes, who are clinically diagnosed with neonatal convulsions. Exclusion criteria include infants older than 30 days or those with movement disorders that mimic seizures, such as jitteriness, benign neonatal sleep myoclonus, hyperekplexia, motor automatisms, or Sandifer syndrome.

After obtaining informed consent from parents or caregivers, enrolled neonates will undergo a comprehensive assessment that includes detailed maternal and perinatal history, physical examination, neurological evaluation, and documentation of seizure semiology. Laboratory investigations include complete blood count, renal and liver function tests, serum electrolytes, blood glucose, metabolic screening when indicated, and infection workup. Neuroimaging such as cranial ultrasound, CT scan, or MRI will be performed based on clinical indications. Additional investigations such as EEG may be used as available.

The primary outcome is to determine the rate of neonatal convulsions among NICU admissions. Secondary outcomes include identification of the most common etiologies, description of clinical patterns, response to treatment, and early in-hospital outcomes such as seizure control, complications, and duration of NICU stay.

Data will be analyzed using standard statistical methods to generate descriptive and analytic comparisons. Findings from this study are expected to fill important knowledge gaps in the local epidemiology of neonatal convulsions and provide evidence to improve diagnostic strategies, early intervention, and quality of neonatal care.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 0 to 30day.
* Children diagnosed with neonatal seizures
* All newborn fullterm,preterm.males and females with neonatal convulsions.

Exclusion Criteria:

* Children above age of 30 day and those with mimic condition as
* jitteriness, benign neonatal sleep myoclonus, motor automatisms,
* hyperekplexia, and Sandifer syndrome..

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population includes neonates aged 0 to 30 days admitted to the Neonatal Intensive Care Unit (NICU) at Assiut University Children's Hospital who are diagnosed with neonatal convulsions. Both full-term and preterm infants of either sex will be included. Neonates with conditions mimicking seizures (e.g., jitteriness, benign neonatal sleep myoclonus, motor automatisms, hyperekplexia, Sandifer syndrome) will be excluded. The target population is expected to be representative of neonates admitted to the NICU with convulsions during the study period from March 2024 to August 2025.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of neonatal convulsions in newborns admitted to the NICU | During NICU stay (up to 30 days of age)
  The proportion of neonates diagnosed with convulsions confirmed clinically and by EEG during hospitalization in the neonatal intensive care unit.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Beniczky S, Tatum WO, Blumenfeld H, Stefan H, Mani J, Maillard L, Fahoum F, Vinayan KP, Mayor LC, Vlachou M, Seeck M, Ryvlin P, Kahane P. Seizure semiology: ILAE glossary of terms and their significance. Epileptic Disord. 2022 Jun 1;24(3):447-495. doi: 10.1684/epd.2022.1430. PMID 35770761
- [Result] Specchio N, Wirrell EC, Scheffer IE, Nabbout R, Riney K, Samia P, Guerreiro M, Gwer S, Zuberi SM, Wilmshurst JM, Yozawitz E, Pressler R, Hirsch E, Wiebe S, Cross HJ, Perucca E, Moshe SL, Tinuper P, Auvin S. International League Against Epilepsy classification and definition of epilepsy syndromes with onset in childhood: Position paper by the ILAE Task Force on Nosology and Definitions. Epilepsia. 2022 Jun;63(6):1398-1442. doi: 10.1111/epi.17241. Epub 2022 May 3. PMID 35503717
- [Result] Kim EH, Shin J, Lee BK. Neonatal seizures: diagnostic updates based on new definition and classification. Clin Exp Pediatr. 2022 Aug;65(8):387-397. doi: 10.3345/cep.2021.01361. Epub 2022 Apr 4. PMID 35381171
- [Result] Shellhaas RA. Neonatal seizures reach the mainstream: The ILAE classification of seizures in the neonate. Epilepsia. 2021 Mar;62(3):629-631. doi: 10.1111/epi.16857. Epub 2021 Feb 26. No abstract available. PMID 33634848